CLINICAL TRIAL: NCT05246917
Title: Rct in croHn's Disease: Comparing mANual (End to End and Kono-s) Versus stapleD Side TO Side Ileocolic Anastomosis (HANDTOEND)
Brief Title: Comparing Manual Versus Stapled Side to Side Ileocolic Anastomosis in Crohn's Disease
Acronym: HAND2END
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Vittoria Bellato, Principal Investigator, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5.2
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Crohn Disease; IBD; Ileocolitis; Crohn's Ileocolitis
Keywords: Recurrence IBD; IBD; Endoscopic Recurrence; Rurgeers Score; Surgical recurrence; Crohn's Ileocolitis; Ileocolic Anastomosis; Crohn's disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: Randomised superiority study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Handsewn ileocolic anastomosis (Experimental): Randomised comparison of handsewn (end-to-end and the Kono-S) with the side-to-side stapled anastomosis.
  to use a manual anastomosis technique avoiding stapled technique to verify if stapled anastomosis can cause ulcers at endoscopic follow up with systematic overscoring
  Interventions: Procedure: Handsewn anastomosis
- Side to side stapled anastomosis (No Intervention): Randomised comparison of handsewn (end-to-end and the Kono-S) with the side-to-side stapled anastomosis.
  to use a manual anastomosis technique avoiding stapled technique to verify if stapled anastomosis can cause ulcers at endoscopic follow up with systematic overscoring

INTERVENTIONS:
Procedure: Handsewn anastomosis — To perform hand sewn anastomosis (either end to end or Kono-s) during the reconstruction face of ileocolic resection
  Arms: Handsewn ileocolic anastomosis

SUMMARY:
RESEARCH QUESTION Are handsewn (end to end and Kono S side to side) anastomoses superior to side to side stapled anastomosis after ileocolic resection for Crohn's disease with respect to endoscopic recurrence, gastrointestinal function and costs.

HYPOTHESIS Stapled side anastomosis advised in ECCO guidelines heal with ulcerations on the staple line causing systematic over scoring of endoscopic recurrence leading to unjustified restarting of expensive drugs reducing QOL and increasing costs. Side to side saccular configuration causes stasis affecting recurrence and dysfunction.

DESIGN Randomised superiority study

POPULATION Patients with Crohn requiring (re)resection of the (neo)terminal ileum

INTERVENTION Kono S and end to end hand sewn anastomosis

USUAL CARE Side to side stapled anastomosis

OUTCOME Endoscopic recurrence (local and central reading) at 6 months

SAMPLE 25% reduction in 2:1 ratio -> 126 + 63 = 189 patients

KEYWORDS Crohn, ileocolic resection, recurrence

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged >18 years
* Ileocolic disease or disease of the neoterminal ileum with an indication for resection
* Concurrent therapies with corticosteroids, 5-ASA drugs, thiopurines, MTX, antibiotics, and anti-TNF therapy are permitted.
* All patients should have undergone a colonoscopy and MR enterography (or CT enterography if MR contraindicated) in last 3 months to assess extent of disease.
* Ability to comply with protocol.
* Competent and able to provide written informed consent.
* Patient must have been discussed in the local MDT

Exclusion Criteria:

* Inability to give informed consent.
* Patients less than 16 years of age.
* Patients undergoing repeated ileocolic resection.
* History of cancer < 5 years which might influence patients prognosis
* Emergent operation. Pregnant or breast feeding.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
6 months endoscopic recurrence of endoscopy using the modified Rutgeerts classification. | 6 months
  The comparison of 6 months endoscopic recurrence between local and central reading of recordings of endoscopy using the modified Rutgeerts classification.

SECONDARY OUTCOMES:
Morbidity | 1 year
  postoperative morbidity measure
Clinical Recurrence | 1 year
  Clinical and surgical recurrence using Clavien Dindo
Inflammatory Bowel Disease Questionnaire (IBDQ) | 1 year
  Quality of life measured with IBD questionnaire
Hospital Costs | 1 year
  Hospital costs per patient in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- irccs San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haanappel AEG, Bellato V, Buskens CJ, Armuzzi A, van der Bilt JDW, de Boer NKH, Danese S, van der Does de Willebois EML, Duijvestein M, van der Horst D, Pellino G, Richir MC, Selvaggi F, Spinelli A, Vignali A, Rosati R, Bemelman WA. Optimising surgical anastomosis in ileocolic resection for Crohn's disease with respect to recurrence and functionality: two international parallel randomized controlled trials comparing handsewn (END-to-end or Kono-S) to stapled anastomosis (HAND2END and the End2End STUDIES). BMC Surg. 2024 Feb 26;24(1):71. doi: 10.1186/s12893-024-02340-3. PMID 38408943